CLINICAL TRIAL: NCT06566872
Title: Collecting Recorded Videos of Colonoscopy Gastroscopy Tests for the Evaluation of the Magentiq Eye Automatic Polyp Detection System (ME-APDS) Medical Device
Brief Title: Collecting Recorded Videos of Colonoscopy and Gastroscopy Tests for the Evaluation of the (ME-APDS).
Status: Recruiting | Type: Observational
Sponsor: Magentiq Eye LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-0041
Record Dates: First submitted 2024-07-14; First posted 2024-08-22 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-07

CONDITIONS: Colon Polyp
Keywords: Polyps
MeSH Terms: conditions — Colonic Polyps; Polyps | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Device: ME-APDS — No Intervention
  Other Names: Automatic Polyp Detection System (ME-APDS) Medical Device

SUMMARY:
The study shall mainly help to better evaluate the performance the ME-APDS device and secondly it may help the development of additional future versions of the ME-APDS.

Primary endpoints

* Clear video of the colon or the stomach or the esophagus achieved during the test.
* Acceptable colon or gastro test performance according to the standards, criteria, and regulations of the medical center of the trial.

Secondary endpoints

• A recorded video of at least 80% of the actual test duration.

DETAILED DESCRIPTION:
Primary objectives • To support the offline evaluation, in objective way, of the performance of the ME-APDS device by testing the sensitivity and specificity and additional statistical parameters of its results achieved from running it on the collected recorded videos of Colonoscopy and Gastroscopy tests of the general population.

Secondary objectives

• Some of the data might be used also for the development of future versions of the ME-APDS

Each subject will pass regular colonoscopy and/or gastroscopy test during which an external recording system connected to the secondary "video out" connector of the endoscopy processing device will record the video presented on the endoscopy device screen from the beginning of the test till its end. The standard off-the shelf recording device will be connected to the endoscopy device's connector by the testing physician or his/her assistant during the test's preparation phase. At the beginning of the test the testing physician or his/her assistant will press on recording start button, and at end of the test, the testing physician or his/her assistant will press on recording stop button. At the end of each week, the recorded video will be backed-up from the recording device to an external storage with two copies, one for record keeping of the main investigator, and one for the sponsoring entity.

Pathology and procedure reports without any identification details will sent to the sponsor with the recorded video.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the - criteria related to regular colonoscopy and/or gastroscopy according to the standard of care at the Gastroenterolgy Department of the selected center, _In addition the following - criteria have to be met to be eligible for the study:

1. Able to read, understand and provide written Informed Consent;
2. Females or males - older than 18 years old

Exclusion Criteria:

Any of the following colonoscopy/gastroscopy related exclusion criteria will exclude the subject from the study:

* Bleeding disorder or unacceptable risk of bleeding
* Terminal illness or life threatening malignancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects shall be recruited by the investigator from within the investigator's patient population of colonoscopy and Gastroscopy. In this study one site will participate and enroll not less than 250 patients and up to 700 subjects according to the inclusion/exclusion criteria. Each subject (not less than 250 patients and up to 700 subjects) included will pass one regular colonoscopy and/or gastroscopy test which will be recorded in the way which is described above.
  Enrolled subjects that did not complete the full course of the study will be replaced.
  Eligibility Each subject will be evaluated by the Investigator to assess his/ her suitability for entry into this study according to the Inclusion and Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To support the offline evaluation, in objective way, of the performance of the ME-APDS device by testing the sensitivity and specificity and additional statistical parameters. | during colonoscopy and gastroscopy procedure
  Clear video of the colon or the stomach or the esophagus achieved during the test.
Acceptable colon or gastro test performance according to the standards, criteria, and regulations of the medical center of the trial. | during colonoscopy and gastroscopy procedure
  Acceptable colon or gastro test performance according to the standards, criteria, and regulations of the medical center of the trial.

SECONDARY OUTCOMES:
A recorded video of at least 80% of the actual test duration. | during colonoscopy and gastroscopy procedure
  A recorded video of at least 80% of the actual test duration.

CONTACTS AND LOCATIONS:
Overall Officials: Haim Shirin, Prof., Principal Investigator — Gastroenterology Department of Shamir Medical Center, Israel
Locations (1):
- Department of Gastroenterology, Shamir Medical Center, Israel, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No